CLINICAL TRIAL: NCT05032261
Title: Norepinephrine Load and Relationship With Prognosis in Critically Patients With Circulatory Shock
Brief Title: ICU Norepinephrine Load
Acronym: ICU_NE_LOAD
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2021/DC-01
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Circulatory Collapse and Shock
Keywords: Norepinephrine load dose; vasopressor dose intensity; vasopressor exposure
MeSH Terms: conditions — Shock | interventions — Norepinephrine; Intensive Care Units

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: surviving Patients: Patients surviving within 5 days of the date of ICU admission for circulatory shock and receiving norepinephrine
  Interventions: Drug: Circulatory shock with norepinephrine in ICU
- Group 2: Deceased patients: Patients deceased within 5 days of the date of ICU admission for circulatory shock and receiving norepinephrine
  Interventions: Drug: Circulatory shock with norepinephrine in ICU

INTERVENTIONS:
Drug: Circulatory shock with norepinephrine in ICU — Circulatory shock with norepinephrine in ICU

SUMMARY:
Norepinephrine is recommended as first-line vasopressor in critically ill patients, regardless of shock etiology. Its advantages over dopamine and/or epinephrine have been demonstrated, especially by reducing tachycardia events. The current guidelines recommend a mean arterial pressure of at least 65 mmHg that in the resuscitation from sepsis-induced hypoperfusion. Some study reported that delay in initiation of vasopressor therapy was associated with an increase mortality risk in patient with septic shock .The recent experts' opinion suggest that " vasopressors should be started early, before (complete) completion of fluid ressuscitation ".

In the event of refractory septic shock, high-dose vasopressors may be used. The precise maximal dose of norepinephrine associated with mortality excess has been poorly studied. High doses have been defined by a cutoff value ranging from 0.5 μg/kg/min to 2 μg/kg/min and recently by 1 μg/kg/min for mortality at 90% and by 0,75 μg/kg/min for mortality at 60%. Furthermore, an increasing vasopressor dosing intensity during the first 24 hours after shock septic was associated with increased mortality depending of fluid administration. If a threshold value of norepinephrine score can be obtained, it could indicate the association with another vasopressor such as vasopressin or surrogates.

The primary aim of the present study aimed to confirm if a given norepinephrine dose is associated with mortality. The secondary aims were the link between mortality and norepinephrine duration, cumulative dose in order to build a score that predicts a futility of increasing norepinephrine dose.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* circulatory shock and admitted in ICU
* with norepinephrine

Exclusion Criteria : Patient without norepinephrine or missing data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with circulatory shock admitted in intensive care unit (ICU) and receiving norepinephrine. All patients older than 18 years recorded between January 1, 2015 and December 31, 2019 were included. Patients with circulatory shock without norepinephrine were excluded.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | Day 5
  Mortality within 5 days of the date of ICU admission for circulatory shock according to norepinephrine intensity

SECONDARY OUTCOMES:
Intensity | Day 5
  Intensity mortality relationship according to norepinephrine duration
Time/Dose Ratio | Day 5
  ratio between time of use and cumulative dose
Norepinephrine dose | Day 5
  score of increasing norepinephrine dose

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Muller, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France

REFERENCES:
- [Result] Ceausu D, Boulet N, Roger C, Alonso S, Lefrant JY, Boisson C, Mura T, Muller L. CRITICAL NOREPINEPHRINE DOSE TO PREDICT EARLY MORTALITY DURING CIRCULATORY SHOCK IN INTENSIVE CARE: A RETROSPECTIVE STUDY IN 3423 ICU PATIENTS OVER 4-YEAR PERIOD. Shock. 2024 Nov 1;62(5):682-687. doi: 10.1097/SHK.0000000000002454. Epub 2024 Aug 28. PMID 39193888